CLINICAL TRIAL: NCT01308593
Title: Investigation Into Brow Aesthetics Using Botox in Conjunction With Juvederm Ultra XC as Evaluated by Patient Satisfaction
Brief Title: Brow Enhancement Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Skin Care and Laser Physicians of Beverly Hills (Other)
Responsible Party: Principal Investigator, Derek H. Jones, M.D., Principal Investigator, Skin Care and Laser Physicians of Beverly Hills
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Brow Study 25856/1
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Brow Ptosis
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Juvederm XC (Active Comparator): Juvederm XC
  Interventions: Device: Juvederm XC
- Botox (Active Comparator): Medication used to block neuromuscular transmission
  Interventions: Drug: Botox

INTERVENTIONS:
Device: Juvederm XC — Filler
  Arms: Juvederm XC
Drug: Botox — 26 units dosed one time
  Arms: Botox

SUMMARY:
Investigation into brow aesthetics using Botox in Conjunction with Juvederm XC as evaluated by patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Men and women

Exclusion Criteria:

* Persons who have not had Botox for months.
* Women who are pregnant, breastfeeding, or trying to get pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Participant satisfaction with combined injection with Botox and Juvederm XC | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Care and Laser Physicians of Beverly Hills, Los Angeles, California, United States